CLINICAL TRIAL: NCT04793932
Title: A Randomized Phase III Trial of Short-course Versus Long-course Pre-operative Chemotherapy With mFOLFIRINOX or PAXG Regimen for Stage I-III Pancreatic Ductal Adenocarcinoma (PDAC)
Brief Title: Short-course Versus Long-course Pre-operative Chemotherapy With mFOLFIRINOX or PAXG (CASSANDRA TRIAL)
Acronym: CASSANDRA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Associazione Italiana per lo Studio del Pancreas (Other)
Collaborators: High Research srl (Unknown); Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PACT21
Record Dates: First submitted 2021-02-28; First posted 2021-03-11 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Pancreas Ductal Adenocarcinoma
Keywords: neoadjuvant chemotherapy; PAXG; mFOLFIRINOX; resectable; borderline resectable

STUDY DESIGN:
Intervention Model Description: 2 by 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PAXG Arm A (Active Comparator): cisplatin 30 mg/m2 every 2 weeks, nab-paclitaxel 150 mg/m2 every 2 weeks, gemcitabine 800 mg/m2 every 2 weeks, capecitabine 1250 mg/m2/day (for 28 consecutive days) in 28-day cycles administered for 4 cycles (4 months).
  Interventions: Drug: PAXG
- mFOLFIRINOX Arm B (Active Comparator): irinotecan 150 mg/m2 day 1, oxaliplatin 85 mg/m2 day 1, folinic acid at a fixed dose of 400 mg/m2, fluorouracil continuous IV infusion 2.4 g/m2 over 46 hours in 14-day cycles administered for 8 cycles (4 months).
  Interventions: Drug: mFOLFIRINOX
- short-course chemotherapy (Active Comparator): Allocated by second randomization after 4 months of chemotherapy to receive immediate surgery followed by 2 further months of the same chemotherapy
  Interventions: Drug: short-course chemotherapy
- long-course chemotherapy (Active Comparator): Allocated by second randomization after 4 months of chemotherapy to receive 2 further months of the same chemotherapy followed by surgery
  Interventions: Drug: long-course chemotherapy

INTERVENTIONS:
Drug: PAXG — Nab-paclitaxel, cisplatin and gemcitabine drugs will be administered on day 1 and 15 every 28 days. Capecitabine tablets will be taken orally on days 1 to 28, every 28 days
  Arms: PAXG Arm A
Drug: mFOLFIRINOX — Oxaliplatin, folinic acid, irinotecan and 5-Fluoruracil will be administered on day 1 and 15 every 28 days
  Arms: mFOLFIRINOX Arm B
Drug: short-course chemotherapy — other two months of chemotherapy after surgery
  Arms: short-course chemotherapy
Drug: long-course chemotherapy — other two months of chemotherapy before surgery
  Arms: long-course chemotherapy

SUMMARY:
The main aim of this study is to compare the efficacy of short-course versus long-course pre-operative chemotherapy with PAXG or mFOLFIRINOX in patients who receive a diagnosis of pancreatic ductal adenocarcinoma (PDAC) resectable or borderline resectable.

DETAILED DESCRIPTION:
Pancreatic cancer is the seventh cause of death in cancer patients and more than 94% of affected patients die of cancer disease. In the majority of cases, the diagnosis is done at an advanced stage and only 10-20% of patients can be treated with a surgical resection. For this neoplasia, a radical resection may be an effective treatment. Nevertheless, results obtained with surgery alone are rather inadequate, showing a median survival of 12-14 months and 2-year survival of almost 20%: it seems evident the necessity to use complementary treatments in order to improve survival rate in this group of patients.

Pancreatic cancer can relapse locally, at the level of tumoral bed, of the regional lymph nodes, on the immediately adjacent peritoneal surface or on contiguous organs. Also, distant metastases are quite frequent, mainly to the liver, at the entire peritoneal surface and, rarely, to the extra-abdominal organs. The rapid appearance of these metastases after surgical resection strongly suggests the presence of subclinical metastatic diffusion at an early phase of the disease.

Currently, combination chemotherapy based on the mFOLFIRINOX regimen is considered the therapeutic standard in the adjuvant setting, in young and fit patients. Unfortunately, mFOLFIRINOX is burdened with strong haematological and extra-haematologic toxicity and just 2/3 of patients are able to complete the treatment. Recently, PAXG regimen [(Cisplatin (P), Abraxane (A), Capecitabine (X), Gemcitabine (G)] when compared to AG in randomized studies, showed an improvement in terms of progression-free survival (PFS) and overall survival in borderline resectable, locally advanced and metastatic patients. To date, several ongoing randomized trials are investigating the efficacy of perioperative or neoadjuvant strategies in early stage PDAC. Only few studies are available regarding neoadjuvant treatment: some are outdated, numerically inconsistent, retrospective, or not randomized. In this scenario, it aims to better investigate pre-operative therapeutic strategy.

For this purpose, two randomizations are planned.

1. FIRST RANDOMIZATION. Eligible patients will be randomized (1:1), stratifying by basal CA19.9 level (<5 ULN vs ≥ 5ULN) and centre to receive:

   PAXG or mFOLFIRINOX for 4 months
2. SECOND RANDOMIZATION. Patients without progression or limiting toxicity after 4 months of the assigned chemotherapy in the study, will be randomized (1:1), stratifying by treatment assigned by the first randomization, to receive 2 further months of the same chemotherapy either BEFORE or AFTER surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Cyto/histological diagnosis of pancreatic ductal adenocarcinoma*;
2. Clinical stage I-III disease according to TNM 8th Ed. 2017 [appendix 1];
3. Resectable or borderline resectable disease, as anatomically defined according to NCCN Guidelines Version 1.2020 - Pancreatic Adenocarcinoma [appendix 2] and biologically defined according to the International consensus on definition and criteria of borderline resectable pancreatic ductal adenocarcinoma 2017 (CA 19.9 > 500 IU/ml) (Isaji et al., 2018);
4. Karnofsky Performance Status > 60% [appendix 3];
5. Age > 18 and ≤ 75 years;
6. Adequate bone marrow function (GB ≥ 3500/mm3, neutrophils ≥1500/mm3, platelets ≥ 100000/mm3, Hb ≥10 g/dl);
7. Adequate kidney function (serum creatinine < 1.5 mg/dL);
8. Adequate liver function:

   * ALT and AST < 3 ULN
   * Serum total bilirubin ≤ 1.5 ULN or in subjects with biliary stenting ≤ 2 ULN;
9. No prior treatment (chemotherapy, radiotherapy and/or surgery) for pancreatic cancer;
10. Women must not be on pregnancy or lactation;
11. Patient of child-bearing potential must agree to use two medically acceptable methods of contraception (one for the patient and one for the partner) during the study and for a minimum of the following 6 months; this applies to patients of both sexes. [appendix 4];
12. Patient information and signed written informed consent.

Exclusion Criteria:

1. Other types of non-ductal tumor of the pancreas, including endocrine tumors or acinar cell adenocarcinoma, cystadenocarcinoma and other periampullary malignancies.
2. Prior (within 1 year) or concurrent malignancies at other sites with the exception of surgically cured carcinoma in-situ of the cervix and basal or squamous cell carcinoma of the skin
3. Symptomatic duodenal stenosis;
4. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment
5. Known infection with hepatitis B or C, or history of human immunodeficiency virus (HIV) infection, or subject receiving immunosuppressive or myelosuppressive medications that would in the opinion of the investigator, increase the risk of serious neutropenic complications
6. Clinical stage IV (including ascites or malignant pleural effusion) disease according to TNM 8th Ed. 2017 [appendix 1];
7. Locally advanced disease according to NCCN Guidelines Version 1.2020 - Pancreatic Adenocarcinoma [appendix 2];
8. Serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the subject's safety or the study data integrity. These include, but are not limited to:

   1. History of connective tissue disorders (eg, lupus, scleroderma, arteritis nodosa)
   2. History of interstitial lung disease, slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies
   3. History of the following within 6 months prior to Cycle 1 Day 1: a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or ECG abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder
9. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
10. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
11. Any condition that confounds the ability to interpret data from the study
12. Any familiar, sociologic or geographic conditions that can potentially interfere with the adhesion to the protocol or to the follow-up;
13. Pre-existing neuropathy
14. c.1679GG, c.1905+1AA, c.2846TT mutations in homozygous in DPYD gene. Dose modification according to DPYD and UGT1A1 mutations are reported in Table 1 (https://www.aiom.it/wp-content/uploads/2019/10/2019_Racc-analisi-farmacogenetiche.pdf.)
15. Inflammatory disease of the colon or rectum, or occlusion or sub-occlusion of the intestine.
16. Concurrent treatment with other experimental drugs;
17. Fructose intolerance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 12 weeks
  to compare in terms of event free survival (EFS) the efficacy of PAXG to that of mFOLFIRINOX. EFS is defined as the time from randomization to: RECIST 1.1 progression [At least a 20 percent increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20 percent, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression]; CA19.9 failure (defined as 2 consecutive increases of serum level ≥20 percent, separated by at least 4 weeks); recurrence; preoperative or intraoperative unresectability; intraoperative evidence of metastases; death for any cause; whichever occurs first. R1 resections will NOT be considered as events whereas R2 resections will be.
Event-free survival | 12 weeks
  to compare in terms of event free survival (EFS) the efficacy of 4 months pre-operative and 2 months postoperative chemotherapy to that of 6 months of pre-operative chemotherapy . EFS is defined as the time from randomization to: RECIST 1.1 progression [At least a 20 percent increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20 percent, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression]; CA19.9 failure (defined as 2 consecutive increases of serum level ≥20 percent, separated by at least 4 weeks); recurrence; preoperative or intraoperative unresectability; intraoperative evidence of metastases; death for any cause; whichever occurs first. R1 resections will NOT be considered as events whereas R2 resections will be.

SECONDARY OUTCOMES:
Overall survival | 36 months
  the time between the date of the patient's enrollment and the death of the patient for any cause or the last time the patient was seen alive
RECIST 1.1 radiological response | 4-6 months
  Radiological response evaluation during the treatment by using RECIST 1.1 criteria
Ca19.9 response rate | 4-6 months
  Biochemical response evaluation during the treatment by using this specific marker
Surgery outcome | 4-6 months after chemotherapy
  The evaluation of resectability rate.
Surgery outcome | 4-6 months after chemotherapy
  The evaluation of surgical mortality and morbidity rate.
Surgery outcome | 4-6 months after chemotherapy
  The evaluation of intra- and post-operative metastasis rate.
Surgery outcome | 4-6 months after chemotherapy
  The evaluation of N0 and R0 resections rate.
Incidence of Treatment Adverse Events | 4-6 months
  The evaluation of drugs safety and tolerability by SAE report
Quality of life | 4-6 months
  Impact of treatment on quality of life assessed by the latest version of the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30)
Quality of life | 4-6 months
  Impact of treatment on quality of life assessed by the European Organization for Research and Treatment of Cancer Quality of Life scale for pancreatic cancer (EORTC QLQ - PAN26)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Reni, MD, Study Chair — IRCCS San Raffaele
Locations (22):
- Italy (22):
  - Oncologia Medica e Prevenzione Oncologica Centro di riferimento oncologico (CRO), IRCCS, Aviano
  - Oncologia Medica Az. Ospedaliera Istituto Tumori "Giovanni Paolo II", Bari
  - Oncologia ASST pg23, Bergamo
  - Oncologia Medica Azienda Universitaria Ospedaliera Policlinico Sant'Orsola-Malpighi, Bologna
  - Oncologia Medica dell'Az.Ospedaliera Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Oncologia Medica AOU Careggi, Florence
  - Oncologia Ospedale Generale Provinciale, Macerata
  - Oncologia Medica dell'Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Oncologia dell'Istituto Clinico Humanitas, Milan
  - IRCCS San Raffaele, Milan
  - Oncologia Medica Falck Niguarda, Milan
  - Oncologia Medica Az Ospedaliera AOU Cagliari Policlinico Universitario Dullio Casula, Monserrato
  - Oncologia Medica AOU FEDERICO II, Naples
  - Oncologia Medica 1 Ospedaliera Istituto Oncologico Veneto IRCCS, Padua
  - Oncologia Medica Arnas Civico, Palermo
  - Oncologia Medica 2 Az. Ospedaliera Universitaria Pisana, Pisa
  - Oncologia Medica Az. Ospedaliera Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome
  - Chirurgia Generale e Oncologica dell'AZ. Ospedaliera Ordine Mauriziano, Torino
  - Divisione Chirurgica Az. Ospedaliera AULSS2, Treviso
  - SOC di Oncologia Az. Ospedaliera Sanitaria Universitaria Friuli Centrale-P.O. "S. Maria della Misericordia", Udine
  - Chirurgia generale e del Pancreas Azienda Ospedaliera Universitaria Integrata, Verona
  - Oncologia ULSS8 Berica, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reni M, Cereda S, Mazza E, Passoni P, Nicoletti R, Balzano G, Zerbi A, Arcidiacono PG, Staudacher C, Di Carlo V. PEFG (cisplatin, epirubicin, 5-fluorouracil, gemcitabine) regimen as second-line therapy in patients with progressive or recurrent pancreatic cancer after gemcitabine-containing chemotherapy. Am J Clin Oncol. 2008 Apr;31(2):145-50. doi: 10.1097/COC.0b013e31814688f7. PMID 18391598
- [Background] Reni M, Balzano G, Aprile G, Cereda S, Passoni P, Zerbi A, Tronconi MC, Milandri C, Saletti P, Rognone A, Fugazza C, Magli A, Di Muzio N, Di Carlo V, Villa E. Adjuvant PEFG (cisplatin, epirubicin, 5-fluorouracil, gemcitabine) or gemcitabine followed by chemoradiation in pancreatic cancer: a randomized phase II trial. Ann Surg Oncol. 2012 Jul;19(7):2256-63. doi: 10.1245/s10434-011-2205-2. Epub 2012 Jan 12. PMID 22237835
- [Background] Reni M, Balzano G, Zanon S, Passoni P, Nicoletti R, Arcidiacono PG, Pepe G, Doglioni C, Fugazza C, Ceraulo D, Falconi M, Gianni L. Phase 1B trial of Nab-paclitaxel plus gemcitabine, capecitabine, and cisplatin (PAXG regimen) in patients with unresectable or borderline resectable pancreatic adenocarcinoma. Br J Cancer. 2016 Jul 26;115(3):290-6. doi: 10.1038/bjc.2016.209. Epub 2016 Jul 12. PMID 27404453
- [Background] Reni M, Balzano G, Zanon S, Zerbi A, Rimassa L, Castoldi R, Pinelli D, Mosconi S, Doglioni C, Chiaravalli M, Pircher C, Arcidiacono PG, Torri V, Maggiora P, Ceraulo D, Falconi M, Gianni L. Safety and efficacy of preoperative or postoperative chemotherapy for resectable pancreatic adenocarcinoma (PACT-15): a randomised, open-label, phase 2-3 trial. Lancet Gastroenterol Hepatol. 2018 Jun;3(6):413-423. doi: 10.1016/S2468-1253(18)30081-5. Epub 2018 Apr 4. PMID 29625841
- [Background] Reni M, Zanon S, Balzano G, Passoni P, Pircher C, Chiaravalli M, Fugazza C, Ceraulo D, Nicoletti R, Arcidiacono PG, Macchini M, Peretti U, Castoldi R, Doglioni C, Falconi M, Partelli S, Gianni L. A randomised phase 2 trial of nab-paclitaxel plus gemcitabine with or without capecitabine and cisplatin in locally advanced or borderline resectable pancreatic adenocarcinoma. Eur J Cancer. 2018 Oct;102:95-102. doi: 10.1016/j.ejca.2018.07.007. Epub 2018 Aug 24. PMID 30149366
- [Background] Reni M, Zanon S, Peretti U, Chiaravalli M, Barone D, Pircher C, Balzano G, Macchini M, Romi S, Gritti E, Mazza E, Nicoletti R, Doglioni C, Falconi M, Gianni L. Nab-paclitaxel plus gemcitabine with or without capecitabine and cisplatin in metastatic pancreatic adenocarcinoma (PACT-19): a randomised phase 2 trial. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):691-697. doi: 10.1016/S2468-1253(18)30196-1. Epub 2018 Jul 7. PMID 30220407
- [Derived] Reni M, Macchini M, Orsi G, Procaccio L, Malleo G, Carconi C, Rapposelli IG, Bencardino K, Scartozzi M, Balzano G, Tamburrino D, Merelli B, Sperti E, Belfiori G, Liscia N, Bozzarelli S, Di Marco M, Tamburini E, Milella M, Lonardi S, Ercolani G, Mazzola M, Palumbo D, Torri V, Falconi M. Preoperative mFOLFIRINOX versus PAXG for stage I-III resectable and borderline resectable pancreatic ductal adenocarcinoma (PACT-21 CASSANDRA): results of the first randomisation analysis of a randomised, open-label, 2 x 2 factorial phase 3 trial. Lancet. 2026 Dec 20;406(10522):2945-2956. doi: 10.1016/S0140-6736(25)01685-X. Epub 2025 Nov 20. PMID 41275879